CLINICAL TRIAL: NCT05670106
Title: A Prospective, Open-label, Multi-center, Single-arm, Phase II Study to Evaluate the Efficacy, Safety, Pharmacokinetics and Dosimetry of [177Lu]Lu-PSMA-617 in Chinese Adult Male Patients With Progressive PSMA-Positive Metastatic Castration-Resistant Prostate Cancer (mCRPC)
Brief Title: A Study to Evaluate the Efficacy, Safety, Pharmacokinetics and Dosimetry of [177Lu]Lu-PSMA-617 in Chinese Adult Male Patients With Progressive PSMA-Positive mCRPC
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAAA617A12201
Record Dates: First submitted 2022-11-07; First posted 2023-01-04 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-10

CONDITIONS: Metastatic Castration-Resistant Prostate Cancer (mCRPC)
Keywords: Chinese adult male population; therapeutic agent lutetium (177Lu) vipivotide tetraxetan; AAA617; [177Lu]Lu-PSMA-617; radiolabeled compound gallium (68Ga) gozetotide; [68Ga]Ga-PSMA-11; Progressive PSMA-Positive Metastatic Castration-Resistant Prostate Cancer; Overall Response Rate; ORR; Prostate-specific Membrane Antigen; PSMA; Taxane; Androgen Receptor Pathway Inhibitor; ARPI
MeSH Terms: interventions — gallium 68 PSMA-11

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- [177Lu]Lu-PSMA-617 plus best supportive/best standard of care (BS/BSOC) (Experimental): Patients will receive the investigational product 7.4 GBq (+/- 10%) 177Lu-PSMA-617 intravenously every 6 weeks (+/- 1 week) for a maximum of 6 cycles. Best supportive/best standard of care (BS/BSOC) may be used
  Interventions: Drug: [177Lu]Lu-PSMA-617; Other: Best supportive/best standard of care (BS/BSOC); Drug: 68Ga-PSMA-11

INTERVENTIONS:
Drug: [177Lu]Lu-PSMA-617 — Administered intravenously once every 6 weeks (1 cycle) for a maximum of 6 cycles.
  Other Names: AAA617
Other: Best supportive/best standard of care (BS/BSOC) — Best supportive/best standard of care as defined by the local investigator
Drug: 68Ga-PSMA-11 — Administered single intravenous dose of approximately 150 MBq. Administered dose could not be lower than 111 MBq or higher than 259 MBq (3 - 7 mCi).

SUMMARY:
The purpose of this study was to assess the efficacy, safety, tolerability, Pharmacokinetic(s) (PK) and dosimetry of [177Lu]Lu-PSMA-617 when administered in addition to Best Supportive/Best Standard of Care (BSC/BSoC) in Chinese participants with progressive PSMA-positive mCRPC who received at least 1 novel androgen receptor pathway inhibitor (ARPI) and were previously treated with 1 to 2 taxane regimens. Furthermore, the safety, PK, and dosimetry of [68Ga]Ga-PSMA-11 were assessed.

Data from this study will be used to bridge global pivotal phase III study (VISION, AAA617A12301) and to support China registration of [177Lu]Lu-PSMA-617 as a novel anticancer modality, namely radioligand therapy, in mCRPC.

DETAILED DESCRIPTION:
This was a 2-part study:

1. Main part: Thirty participants with at least 1 measurable lesion by PCWG3-modified RECIST v1.1 criteria were enrolled in the main part. The primary endpoint of confirmed overall response rate (ORR) was analyzed with participants in this part and was assessed via independent centralized review of radiographic images provided by the Investigator and as outlined in PCWG3-modified RECIST v1.1 criteria.
2. Extension part: The extension part enrolled additional 30 participants with or without measurable lesions following the main part. The secondary endpoints were analyzed with all participants in both main part and extension part.

Screening and enrollment period:

Written informed consent form (ICF) was obtained prior to any screening procedures. All screening procedures described in the Assessment Schedule were completed within 28 days prior to enrollment, except for radiographic imaging assessment, which was done within 21 days prior to enrollment.

The participants were assessed for eligibility and underwent a mandatory [68Ga]Ga-PSMA-11 Positron Emission Tomography (PET)/Computed Tomography (CT) scan to evaluate Prostate-specific Membrane Antigen (PSMA) positivity for eligibility as assessed by central readers. Only participants with PSMA positive cancer and confirmed eligibility criteria were enrolled.

Following completion of all required screening procedures and verifying participant eligibility, the participant was enrolled. [177Lu]Lu-PSMA-617 was ordered in parallel with interactive response technology (IRT) enrollment registration to allow at least 2 weeks to order and deliver [177Lu]Lu-PSMA-617.

Treatment period:

In principle, all participants should begin [177Lu]Lu-PSMA-617 dosing within 14 days after enrollment registration. However, Cycle 1 Day 1 (C1D1) could be delayed by up to an additional 3 days only for unexpected scheduling delays. Participants received 7.4 Gigabecquerel (GBq) (200 Millicuries (mCi)) +/- 10% [177Lu]Lu-PSMA-617 once every 6 weeks for a planned 6 cycles. BSC/BSoC coud be used, including available care for the eligible participants according to best institutional practice. ARPIs (e.,g., abiraterone, etc.) were allowed. BSC/BSoC for each participant was selected at the discretion of the Investigator prior to [177Lu]Lu-PSMA-617 administration, and could be modified over time as needed. BSC/BSoC was administered per the physician's orders according to clinical best practice.

Radiographic imaging (CT with contrast/Magnetic Resonance Imaging (MRI) and bone scan) was done at every 8 weeks (± 4 days) after first dose of [177Lu]Lu-PSMA-617 for the first 24 weeks (independent of dose delays), then every 12 weeks (± 4 days) thereafter and at End of Treatment (EOT) Visit (if not done within 28 days of EOT) until radiographic disease progression confirmed by central reader, death, withdrawal of consent, loss to follow-up, or subject/guardian's decision.

After the last day of study treatment period of [177Lu]Lu-PSMA-617 (i.e. after completion of 6 cycles of treatment OR treatment discontinuation for any reason) [e.g. upon radiographic progression as confirmed by blinded independent centralized review]), the participants have to have an EOT visit performed ≤ 7 days and enter into the Post-treatment Follow-up period.

If a participant withdrew consent for the treatment period of the study, an EOT is supposed to be done and the participant would enter into the Post-treatment Follow-up unless he specifically withdrew consent for post-treatment follow-up.

Post-treatment Follow-up period:

1. 30-day Safety Follow-up. All treated participants are to have a safety follow-up conducted approximately 30 days after EOT visit.
2. Long term Follow-up. The long-term follow-up would start after the 30-day Safety follow-up and would last until study completion. If a participant in the long-term follow-up period discontinued treatment for reasons other than BICR-determined radiographic progression, his tumor assessments were required to be performed every 8 weeks after first dose of study treatment for the first 24 weeks (week 9, 17, 25) and then every 12 weeks (week 37, 49, etc) until confirmation of radiographic progression by BICR. The long-term follow-up period also includes the collection of survival and treatment updates, patient reported outcomes (PROs), serious adverse events (suspected to be related to study treatment), as well as blood sampling for hematology, chemistry testing, coagulation, and PSA. The visits are supposed to be carried out every 12 weeks (± 4 weeks) until death, lost to follow-up, withdrawal of consent, opposition to use data/biological samples or study completion, whichever occurs first. This follow-up allows the data collection on medically significant long-term toxicities, such as long-term radiotoxicity.

If the participant withdrew consent for the collection of blood samples, PROs, and imaging assessments during the long-term follow-up, the information on survival, serious adverse events (SAEs) related to study treatment and post-treatment antineoplastic therapy are to be collected.

PK/dosimetry assessments:

Both PK and dosimetry of [68Ga]Ga-PSMA-11 was to be evaluated in at least 10 and up to 12 participants (at least 6 participants in main part). PK and dosimetry of [68Ga]Ga-PSMA-11 could be evaluated in any participant regardless of his PSMA status.

Both PK and dosimetry of [177Lu]Lu-PSMA-617 are to be evaluated in at least 10 and up to 12 participants (at least 6 participants in main part).

Participants who took part in PK and dosimetry evaluation of [177Lu]Lu-PSMA-617 were to take part in the efficacy and safety evaluation together with the other participants. The treatment and assessment procedure followed the same as above.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent must be obtained before any assessment is performed.
* Participants must be Chinese male adults >= 18 years of age.
* Participants must have histological, pathological, and/or cytological confirmation of prostate cancer.
* Participants must be [68Ga]Ga-PSMA-11 PET/CT scan positive, and eligible as determined by the sponsor's central reader according to the VISION read rules.
* Participants must have a castrate level of serum/plasma testosterone (< 50 ng/dl, or < 1.7 nmol/L).
* Participants must have received at least one ARPI (such as enzalutamide and/orabiraterone).
* Participants must have been previously treated with at least 1, but no more than 2 previous taxane regimens.

  * A taxane regimen is defined as a minimum exposure of 2 cycles of a taxane. If a participant has received only 1 taxane regimen, the participant is eligible if: the participants' physician deems him unsuitable to receive a second taxane regimen (e.g., frailty assessed by geriatric or health status evaluation or intolerance, etc.)
* Documented progressive mCRPC, based on at least 1 of the following criteria:

  * Serum/plasma PSA progression defined as 2 consecutive increases in PSA measured at least 1 week apart, the minimal start value is 2.0 ng/ml
  * Soft-tissue progression defined based on PCWG3-modified RECIST v1.1 (Eisenhauer et al 2009, Scher et al 2016)
  * Progression of bone disease: two new lesions; only positivity on the bone scan defines metastatic disease to bone (PCWG3 criteria (Scher et al 2016)
* Participants must have >= 1 metastatic lesion that is present on baseline CT, MRI or bone scan imaging obtained =< 21 days prior to enrollment via central reading.

  * In main part: participant must have at least one measurable lesion by PCWG3-modified RECIST v1.1 via central reading
* Participants must have adequate organ function:

  * Bone marrow reserve:
  * White blood cell (WBC) count >= 2.5 × 109/L OR absolute neutrophil count (ANC) >= 1.5 × 109/L
  * Platelets >=100 × 109/L
  * Hemoglobin >= 9 g/dL
  * Hepatic:
  * Total bilirubin =< 1.5 x the institutional upper limit of normal (ULN). For participants with known Gilbert's Syndrome =< 3 × ULN is permitted
  * Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) =< 3.0 × ULN OR =< 5.0 × ULN for participants with liver metastases
  * Renal:
  * eGFR >= 50 mL/min/1.73m2 using the Modification of Diet in Renal Disease (MDRD) equation
* Albumin >3.0 g/dL.

Exclusion Criteria:

* Previous treatment with Strontium-89, Samarium-153, Rhenium-186, Rhenium-188, Radium-223 or hemi-body irradiation.
* Previous PSMA-targeted radioligand therapy.
* Any systemic anti-cancer therapy (e.g. chemotherapy, immunotherapy or biological therapy [including monoclonal antibodies], APRI is not included) within 28 days prior to day of enrollment.
* Any investigational agents (e.g. poly adenosine diphosphate-ribosyl polymerase inhibitors [PARPi]) within 28 days prior to day of enrollment.
* History of hypersensitivity to any of the study drugs or its excipients or to drugs of similar chemical classes.
* Other concurrent cytotoxic chemotherapy, immunotherapy, radioligand therapy, or investigational therapy.
* Transfusion for the sole purpose of making a subject eligible for study inclusion.
* Participants with a history of central nervous system (CNS) metastases who are neurologically unstable, symptomatic, or receiving corticosteroids for the purpose of maintaining neurologic integrity.

  * Participants with CNS metastases are eligible if received therapy (surgery, radiotherapy, gamma knife), asymptomatic and neurologically stable without corticosteroids.
  * Participants with epidural disease, canal disease and prior cord involvement are eligible if those areas have been treated, are stable, and not neurologically impaired.
* Symptomatic spinal cord compression, or clinical or radiologic findings indicative of impending cord compression.

Ages: 18 Years to 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Prostate cancer
Enrollment: 62 (Actual)
Dates: Start 2023-05-16 (Actual); Primary Completion 2024-05-17 (Actual); Study Completion 2025-11-14 (Estimated)

PRIMARY OUTCOMES:
Main part: Confirmed Overall Response Rate (ORR) per Blinded Independent Central Review (BICR) | From date of randomization until date of radiographic progression or date of death from any cause, whichever comes first, approx. 1 year
  Confirmed Overall Response Rate (ORR) is defined as the proportion of participants with Best Overall Response (BOR) of Complete Response (CR) or Partial Response (PR). ORR is based on PCWG3-modified RECIST v1.1 response for patients with measurable disease at baseline.

SECONDARY OUTCOMES:
Main & extension parts: Radiographic progression free survival (rPFS) | From date of randomization until date of radiographic progression or date of death from any cause, whichever comes first.
  rPFS is defined as the time (in months) from the date of enrollment to the date of radiographic progression as outlined in PCWG3 guideline or death due to any cause.
Main & extension parts: Overall survival (OS) | From date of randomization until date of death from any cause.
  Overall survival (OS) is defined as the time(in months) from the date of enrollment to the date of death due to any cause. If a participant is not known to have died, then OS will be censored at the latest date the participant was known to be alive (on or before the cut-off date).
Main & extension parts: Overall response rate (ORR) | From date of randomization till radiographic progression or date of death from any cause.
  Overall response rate (ORR)is defined as the proportion of participants with best overall response of complete response or partial response, as per central and local review according to PCWG3 modified RECIST 1.1
Main & extension parts: Disease control rate (DCR) | From date of randomization till radiographic progression or date of death from any cause.
  Disease control rate (DCR) is defined as the proportion of participants with best overall response of complete response or partial response or Stable disease, or non-CR/non-PD, as per central and local review and according to PCWG3-modified RECIST v1.1.
Main & extension parts: Duration of response (DOR) | From date of randomization until date of progression or date of death from any cause.
  Duration of response (DOR) is defined as the time (in months) from the date of the first documented response (CR or PR) to the date of first documented progression according to PCWG3-modified RECIST v1.1 or death due to any cause, among participants with a confirmed response.
Main & extension parts: Time to a first symptomatic skeletal event (TTSSE) | From date of randomization till date of a first SSE or date of death from any cause.
  TTSSE is defined as the time (in months) from the date of enrollment to the date of SSE or death due to any cause. The SSE date is date of the first new symptomatic pathological bone fracture, spinal cord compression, tumor-related orthopedic surgical intervention, requirement for radiation therapy to relieve bone pain, or death due to any cause, whichever comes first.
Main & extension parts: PSA50 response rate | From date of randomization till end of long-term FU.
  PSA response rate is the proportion of PSA responders, defined as a participant who has achieved PSA decrease of >= 50% from baseline that is confirmed by a second consecutive PSA measurement >= 4 weeks later.
Main & extension parts: Progression Free Survival (PFS) | From date of randomization until date of progression or date of death from any cause, whichever come first.
  PFS (Radiographic/clinical/PSA progression) is defined as the time (in months) from the date of enrollment to the date of radiographic, clinical or PSA progression free survival, or death due to any cause, whichever occurs first.
Main & extension parts: European Quality of Life (EuroQol) - 5 Domain 5 Level scale (EQ-5D- 5L) | From date of randomization till the end of long term FU
  FACT-P assesses symptoms/problems related to prostate carcinoma and its treatment. It is a combination of the FACT- General + the Prostate Cancer Subscale (PCS). The FACTGeneral (FACT-G) is a 27 item Quality of Life (QoL) measure that provides a total score as well as subscale scores: Physical (0-28), Functional (0-28), Social (0-28), and Emotional Well-being (0-24). The total score range is between 1-108, higher scores indicates better for total score and subscale scores. PCS is a 12-item prostate cancer subscale that asks about symptoms and problems specific to prostate cancer (Range 0-48, higher scores better). The FACT-P total score is the sum of all 5 subscale scores of the FACT-P questionnaire and ranges from 0-156. Higher scores indicate higher degree of functioning and better quality of life.
Main & extension parts: Functional Assessment of Cancer Therapy - Prostate (FACT-P) Questionnaire | From date of randomization till 30 day safety follow-up or at the end of long term FU for patients prematurely discontinued, assessed up to 57 months (estimated final OS analysis)
  FACT-P assesses symptoms/problems related to prostate carcinoma and its treatment. It is a combination of the FACT- General + the Prostate Cancer Subscale (PCS). The FACTGeneral (FACT-G) is a 27 item Quality of Life (QoL) measure that provides a total score as well as subscale scores: Physical (0-28), Functional (0-28), Social (0-28), and Emotional Well-being (0-24). The total score range is between 1-108, higher scores indicates better for total score and subscale scores. PCS is a 12-item prostate cancer subscale that asks about symptoms and problems specific to prostate cancer (Range 0-48, higher scores better). The FACT-P total score is the sum of all 5 subscale scores of the FACT-P questionnaire and ranges from 0-156. Higher scores indicate higher degree of functioning and better quality of life.
Main & extension parts: Brief Pain Inventory - Short Form (BPI-SF) Questionnaire | From date of randomization till the end of long term FU
  The BPI-SF is a publicly available instrument to assess the pain and includes severity and interference scores. BPI-SF is an 11-item selfreport questionnaire that is designed to assess the severity and impact of pain on daily functions of a participant. Pain severity score is a mean value for BPI-SF questions 3, 4, 5 and 6 (questions inquiring about the extent of pain, where the extent is ranked from 0 [no pain] to 10 [pain as bad as you can imagine]). Pain severity progression is defined as an increase in score of 30% or greater from baseline without decrease in analgesic use.
Main & extension parts: Number of Participants with Treatment Emergent Adverse Events | From day of the first administration of study treatment to 30 days after EOT or to the last [177Lu]Lu-PSMA-617 dose date + 41 days, whichever is later.
  The distribution of adverse events will be done via the analysis of frequencies for treatment emergent Adverse Event (TEAEs) and Serious Adverse Event (TESAEs), through the monitoring of relevant clinical and laboratory safety parameters.
Main & extension parts: Area under the blood concentration-time curve from time zero to the time of last quantifiable concentration (AUClast) of [177Lu]Lu-PSMA-617 | Cycle 1 Week 1(Day 1) and Cycle 1 Week 2(Day 8): Pre dose, 0(End of infusion), 20 & 60 mins(+/- 5 mins), 2 & 4 hours(+/-30 mins), 24 hours(+/- 2 hr), 48 hours(+/- 4 hr), 72 hours(+/- 6 hr), 168 hours(+/- 12 hr) from the end of infusion (1 cycle=42 days)
  Venous whole blood samples will be collected for activity-based pharmacokinetics characterization of [177Lu]Lu-PSMA-617 in at least 10 and up to 14 patients. AUClast will be listed and summarized using descriptive statistics.
Main & extension parts: Observed maximum blood concentration (Cmax) of [177Lu]Lu-PSMA-617 | Cycle 1 Week 1(Day 1) and Cycle 1 Week 2(Day 8): Pre dose, 0(End of infusion), 20 & 60 mins(+/- 5 mins), 2 & 4 hours(+/-30 mins), 24 hours(+/- 2 hr), 48 hours(+/- 4 hr), 72 hours(+/- 6 hr), 168 hours(+/- 12 hr) from the end of infusion (1 cycle=42 days)
  Venous whole blood samples will be collected for activity-based pharmacokinetics characterization of [177Lu]Lu-PSMA-617 in at least 10 and up to 14 patients. Cmax will be listed and summarized using descriptive statistics.
Main & extension parts: Blood concentration of [177Lu]Lu-PSMA-617 | Cycle 1 Week 1(Day 1) and Cycle 1 Week 2(Day 8): Pre dose, 0(End of infusion), 20 & 60 mins(+/- 5 mins), 2 & 4 hours(+/-30 mins), 24 hours(+/- 2 hr), 48 hours(+/- 4 hr), 72 hours(+/- 6 hr), 168 hours(+/- 12 hr) from the end of infusion (1 cycle=42 days)
  Venous whole blood samples will be collected for activity-based pharmacokinetics characterization of [177Lu]Lu-PSMA-617 in at least 10 and up to 14 patients. Blood concentration of [177Lu]Lu-PSMA-617 will be summarized with descriptive statistics.
Main & extension parts: Organ absorbed dose of [177Lu]Lu-PSMA-617 | Cycle 1 Week 1(Day 1) and Cycle 1 Week 2(Day 8): 1~2 & 4 hours, 18~26 hours, 48 hours(+/- 12 hr), 168 hours(+/- 12 hr) from the end of infusion (1 cycle=42 days)
  The quantity of ionizing radiation absorbed by organs and tissues will be summarized with descriptive statistics.
Main & extension parts: Area under the blood concentration-time curve from time zero to the time of last quantifiable concentration (AUClast) of [68Ga]Ga-PSMA-11 | Screening (Day -42 to Day -14) : 5 mins (+/- 3 mins), 15 & 30 & 45 mins (+/- 5 mins), 85 mins (+/- 10 mins), 175 & 245 mins (+/- 30 mins) from the end of infusion
  Venous whole blood samples will be collected for activity-based pharmacokinetics characterization of [68Ga]Ga-PSMA-11 in at least 10 and up to 14 patients. AUClast will be listed and summarized using descriptive statistics.
Main & extension parts: Observed maximum blood concentration (Cmax) of [68Ga]Ga-PSMA-11 | Screening (Day -42 to Day -14) : 5 mins (+/- 3 mins), 15 & 30 & 45 mins (+/- 5 mins), 85 mins (+/- 10 mins), 175 & 245 mins (+/- 30 mins) from the end of infusion
  Venous whole blood samples will be collected for activity-based pharmacokinetics characterization of [68Ga]Ga-PSMA-11 in at least 10 and up to 14 patients. Cmax will be listed and summarized using descriptive statistics.
Main & extension parts: Blood concentration of [68Ga]Ga-PSMA-11 | Screening (Day -42 to Day -14) : 5 mins (+/- 3 mins), 15 & 30 & 45 mins (+/- 5 mins), 85 mins (+/- 10 mins), 175 & 245 mins (+/- 30 mins) from the end of infusion
  Venous whole blood samples will be collected for activity-based pharmacokinetics characterization of [68Ga]Ga-PSMA-11 in at least 10 and up to 14 patients. Blood concentration of [68Ga]Ga-PSMA-11 will be summarized with descriptive statistics.
Main & extension parts: Organ absorbed dose of [68Ga]Ga-PSMA-11 | Screening (Day -42 to Day -14): 30 mins (+/- 5 mins), 60 mins (+/- 10 mins), 120 mins (+/- 20 mins) and 255 mins (+/- 30 mins) from the end of infusion
  The quantity of ionizing radiation absorbed by organs and tissues will be summarized with descriptive statistics.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (10):
- China (10):
  - Novartis Investigative Site, Guangzhou, Guangdong
  - Novartis Investigative Site, Zhengzhou, Henan
  - Novartis Investigative Site, Wuhan, Hubei
  - Novartis Investigative Site, Nanjing, Jiangsu
  - Novartis Investigative Site, Xian, Shanxi
  - Novartis Investigative Site, Chengdu, Sichuan
  - Novartis Investigative Site, Beijing
  - Novartis Investigative Site, Guangzhou
  - Novartis Investigative Site, Shanghai
  - Novartis Investigative Site, Tianjin

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent expert panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data is currently available according to the process described on www.clinicalstudydatarequest.com
URL: https://www.clinicalstudydatarequest.com